CLINICAL TRIAL: NCT01022229
Title: Phase 3 Study of a Compound Natural Health Product in Children With ADHD
Brief Title: The Safety and Efficacy of a Compound Natural Health Product in Children With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Canadian College of Naturopathic Medicine (Other)
Collaborators: Health Canada (Other Government); Centre for Addiction and Mental Health (Other); SickKids Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCNM-0903
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Disorder; Pediatrics; Attention; Impulsivity; Complementary Therapies
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Impulsive Behavior | interventions — Zinc; Magnesium; Vitamin B 6; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Compound Natural Health Product (Experimental): 15 study participants who will receive the compound natural health product.
  Interventions: Dietary Supplement: Compound Natural Health Product
- Placebo (Placebo Comparator): 15 participants will receive placebo natural health product.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Compound Natural Health Product — * 15-35 mg zinc citrate
  * 150-350 mg magnesium lactate
  * 30-70 mg pyridoxine hydrochloride
  * 150-350 mg calcium ascorbate
  Doses are weight based. Chewable tablets are taken 2 times/day with food for the duration of the study
  Other Names: Zinc; Magnesium; Vitamin B6; Vitamin C
  Arms: Compound Natural Health Product
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the use of a natural health product, as compared to placebo (an inactive substance), in managing the symptoms of ADHD. The natural health product contains the nutrients zinc, magnesium, vitamin B6 and vitamin C. Each of these nutrients has some evidence to suggest that children with ADHD might be lacking them. As such, children with ADHD might benefit from supplementing their diets with these nutrients, especially ADHD children who have below average levels.

This study will measure whether the severity of ADHD symptoms is greater in children with low levels of zinc, magnesium, and vitamin B6, and whether the severity of ADHD symptoms will decrease with supplementation of these nutrients. This study will also monitor for any adverse reactions or side effects from taking these nutrients in children.

Although these natural health products are commercially available, the use of them as a supplement or placebo in this study has been approved for use in this study by the Natural Health Products Directorate of Health Canada.

DETAILED DESCRIPTION:
The study is a randomized control, double blinded trial. A population of 30 children diagnosed with ADHD (n=30) will be randomly assigned to the NHP group (n=15) or a placebo group (n=15). The NHP group will be provided with a weight-based dose of a chewable natural health product containing zinc, magnesium, vitamin B6 and vitamin C for 10 weeks, with an additional follow-up post intervention at 20 weeks. The placebo group will be administered a chewable placebo tablet and will follow the same regimen. Severity of ADHD symptoms will be measured at baseline, week 5 and week 10 using the Connor-3 Parent and SNAP-IV validated questionnaires. Nutritional status will be monitored at baseline and week 10 for changes in serum zinc and erythrocyte magnesium. Children will be monitored for any adverse reactions that may occur using the investigational product.Following the informed consent process, participants will undergo a structured psychiatric interview prior to enrollment and will have 4 30 minute study visits and 2 10 minute telephone calls throughout the study. Blood samples will be taken 2 times with the use of a topical anesthetic to decrease sensation during the blood draw. Once enrolled, children can withdraw from the study at any time if assent to participate is withdrawn.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children age 6-12 diagnosed with ADHD of any subtype according to DSM-IV criteria. A structured diagnostic interview (Kiddie Sads Present and Lifetime Version) will be conducted to confirm diagnosis of ADHD and assess for comorbid mental health disorders
* Primary caregiver (parent or guardian) has given informed consent; child participant gives ongoing assent throughout the study.

Exclusion Criteria:

* Changes to participants' ADHD medication within 6 weeks of study onset.
* Diagnosis of additional mental health disorder using the Kiddie Sads.
* Diagnosis of cancer.
* Antibiotic use for periods greater than 2 weeks within the 10 weeks prior to the study
* Diagnosis of Type 1 diabetes and insulin use
* Low serum ferritin/iron deficiency (<30 ng/ml)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2013-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Connors-3 Parent Rating Scale | Baseline, week 5, week 10 and follow-up at week 20

SECONDARY OUTCOMES:
Nutritional status of zinc and magnesium | Week 0 and week 10
Adverse events | Throughout study
SNAP-IV Parent ADHD questionnaire | Week 0, week 5 and week 10

CONTACTS AND LOCATIONS:
Overall Officials: Umesh Jain, MD, Study Director — The Centre for Addiction and Mental Health
Locations (1):
- Robert Schad Naturopathic Clinic, Toronto, Ontario, Canada